CLINICAL TRIAL: NCT02322801
Title: Observational Safety Study of Rituximab in Patients Diagnosed With Rheumatoid Arthritis (RA) Who Did Not Respond Adequately to TNF-alpha Blocker
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21774
Record Dates: First submitted 2014-12-19; First posted 2014-12-23 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multi-center, observational, retrospective-prospective cohort study will investigate the safety of rituximab (MabThera) by collecting data from daily clinical practice on the use of rituximab and its relative clinical impact, particularly with regard to adverse events. Data from each patient will be collected over 24 months after enrolment in the study. Target sample size is up to 325 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with RA who did not respond adequately to anti-TNF-alpha and who started rituximab (RTX) treatment in the 12 months before site initiation and were still under treatment when enrollment starts

Exclusion Criteria:

* Patients with serious infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with RA who did not respond adequately to anti-TNF-alpha
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Percent of patients with at least one grade 3 or 4 adverse event since starting RTX treatment and in the 24 months after study enrollment | Up to 31 months (24 months each patient)

SECONDARY OUTCOMES:
Percent of patients with at least one severe adverse event (SAE) | Up to 31 months (24 months each patient)
Percent of patients who discontinued therapy with RTX | Up to 31 months (24 months each patient)
Time to "re-treatment" with RTX | Up to 31 months (24 months each patient)
Features of responders to RTX therapy in terms of co-morbidity and concomitant drugs | Up to 31 months (24 months each patient)
Time to response and duration of response to RTX | Up to 31 months (24 months each patient)
Percent of patients who achieve remission and relative quality of life (QoL) at 6, 12 and 24 months versus baseline | Up to 31 months (24 months each patient)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (43):
- Italy (43):
  - Pescara, Abruzzo
  - Brindisi, Apulia
  - Martina Franca, Apulia
  - San Cesario di Lecce, Apulia
  - San Daniele Del Friuli, Apulia
  - Mormanno, Calabria
  - Napoli, Campania
  - Scafati, Campania
  - Bologna, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Piacenza, Emilia-Romagna
  - Gorizia, Friuli Venezia Giulia
  - Trieste, Friuli Venezia Giulia
  - Albano Laziale, Lazio
  - Rieti, Lazio
  - Rome, Lazio
  - Viterbo, Lazio
  - Arenzano, Liguria
  - Savona, Liguria
  - Cremona, Lombardy
  - Legnano, Lombardy
  - Milan, Lombardy
  - Monza, Lombardy
  - Rozzano, Lombardy
  - Cuneo, Piedmont
  - Novara, Piedmont
  - Pinerolo, Piedmont
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Monserrato, Sardinia
  - Catania, Sicily
  - Palermo, Sicily
  - Arezzo, Tuscany
  - Florence, Tuscany
  - Massa, Tuscany
  - Pisa, Tuscany
  - Pontedera, Tuscany
  - Prato, Tuscany
  - Treviso, Veneto
  - Valeggio sul Mincio, Veneto
  - Venezia, Veneto
  - Verona, Veneto
  - Vicenza, Veneto